CLINICAL TRIAL: NCT03030235
Title: Effects of Dapagliflozin on Biomarkers, Symptoms and Functional Status in Patients With PRESERVED Ejection Fraction Heart Failure
Brief Title: Dapagliflozin in PRESERVED Ejection Fraction Heart Failure
Acronym: PRESERVED-HF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Saint Luke's Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1690C00053
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Results first posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-09

CONDITIONS: Chronic Heart Failure With Preserved Systolic Function
Keywords: heart failure; dapagliflozin; SGLT-2 inhibitors
MeSH Terms: conditions — Heart Failure | interventions — dapagliflozin; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Active Comparator): Dapagliflozin 10 mg oral tablet, once daily, for 12 weeks
  Interventions: Drug: Dapagliflozin 10Mg Oral Tablet
- Placebo (Placebo Comparator): Dapagliflozin matching placebo oral tablet, once daily, for 12 weeks
  Interventions: Drug: Dapagliflozin matching placebo

INTERVENTIONS:
Drug: Dapagliflozin 10Mg Oral Tablet — Dapagliflozin 10Mg Oral Tablet
  Other Names: Farxiga
  Arms: Dapagliflozin
Drug: Dapagliflozin matching placebo — Dapagliflozin matching placebo
  Other Names: Placebo Oral Tablet
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to evaluate the impact of dapagliflozin, as compared with placebo, on heart failure, disease specific biomarkers, symptoms, health status and quality of life in patients with chronic heart failure with preserved systolic function.

DETAILED DESCRIPTION:
A 12-week randomized, double-blind, placebo-controlled trial to evaluate the effects of once-daily dapagliflozin 10 mg on heart failure disease-specific biomarkers (NTproBNP and BNP), symptoms, health status, and quality of life in patients with chronic heart failure with preserved systolic function. An imaging substudy will also be conducted to explore the effects of dapagliflozin vs. placebo on various echocardiographic parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Symptoms of dyspnea (NYHA class II-IV) without evidence of a non-cardiac or ischemic explanation for dyspnea
2. Ejection fraction (EF) ≥ 45% as determined on imaging study within 24 months of enrolment with no change in clinical status suggesting potential for deterioration in systolic function
3. Elevated NT-proBNP (≥ 225 pg/ml) or BNP (≥ 75 pg/ml). For patients with permanent atrial fibrillation inclusion thresholds will be BNP ≥ 100 pg/mL or NTproBNP ≥ 375 pg/mL
4. Stable medical therapy for heart failure for 15 days as defined by: i. No addition or removal of ACE, angiotensin receptor blockers (ARBs), valsartan/sacubitril, beta-blockers, calcium channel blockers (CCBs) or aldosterone antagonists; ii.No substantial change in dosage (100% or greater increase or decrease from baseline dose) of ACE, ARBs, beta-blockers, CCBs or aldosterone antagonists
5. On a diuretic ≥15 days prior to screening visit and a stable diuretic therapy for 7 days
6. At least one of the following: i. Hospitalization for decompensated HF in the last 12 months; ii. Acute treatment for HF with intravenous loop diuretic or hemofiltration in the last 12 months; iii. Mean pulmonary capillary wedge pressure ≥15 mmHg or LV end diastolic pressure (LVEDP) ≥15 mmHg documented during catheterization at rest, or pulmonary capillary wedge pressure or LVEDP ≥25 mmHg documented during catheterization with exercise; iv. Structural heart disease evidenced by at least one of the following echo findings (any local measurement made within the 24 months prior to screening visit): a) left atrial (LA) enlargement defined by at least one of the following: LA width ≥3.8cm or LA length ≥5.0 cm or LA area ≥20 cm2 or LA volume ≥55 mL or LA volume index ≥29 mL/m2 b) or left ventricular hypertrophy (LVH) defined by septal thickness or posterior wall thickness ≥1.1 cm.

Exclusion Criteria:

1. Decompensated heart failure (hospitalization for heart failure within 7 days prior to screening)
2. History of type 1 diabetes
3. History of diabetic ketoacidosis
4. Estimated glomerular filtration rate (eGFR) < 20 at the screening visit by modified MDRD equation GFR (mL/min/1.73 m2 ) = 175 x (Scr) -1.154 x (Age)-0.203 x (0.742 if female) x (1.210 if African American)
5. Admission for an acute coronary syndrome (ST-elevation MI, non-ST-elevation MI, or unstable angina), percutaneous coronary intervention, or cardiac surgery within 30 days prior to the screening visit.
6. Admission for cardiac resynchronization therapy (CRT) within 90 days prior to the screening visit.
7. Planned cardiovascular revascularization (percutaneous intervention or surgical) or major cardiac surgery (coronary artery bypass grafting, valve replacement, ventricular assist device, cardiac transplantation, or any other surgery requiring thoracotomy, or transcatheter aortic valve replacement) or CRT within the 90 days after the screening visit.
8. Participation in any interventional clinical trial (with an investigational drug or device) that is not an observational registry within 15 days of the screening visit.
9. History of hypersensitivity to dapagliflozin
10. For women of child-bearing potential: Current or planned pregnancy or currently lactating.
11. Life expectancy <1 year at the screening visit
12. Patients who are volume depleted based upon physical examination at the time of the screening or randomization visit
13. BNP <75 pg/mL and NTproBNP<225 pg/mL at the screening visit. For patients with permanent atrial fibrillation exclusion thresholds will be BNP<100 pg/mL and NTproBNP<375pg/mL.
14. Patients currently being treated with any SGLT-2 inhibitor (dapagliflozin, canagliflozin, empagliflozin, ertugliflozin) or having received treatment with any SGLT-2 inhibitor within the 12 weeks prior to the screening visit.
15. Average supine systolic BP <100 mmHg at the screening or randomization visit
16. Current history of bladder cancer
17. Donation of blood or bone marrow 12 weeks prior to the screening visit and no planned donations during the study period
18. Heart failure due to restrictive/infiltrative cardiomyopathy, active myocarditis, constrictive pericarditis, severe stenotic valve disease, and HOCM (hypertrophic obstructive cardiomyopathy).
19. Heart failure due to severe aortic or mitral regurgitation
20. Severe COPD thought to be a primary contributor to dyspnea
21. Isolated right heart failure due to pulmonary disease
22. Active and significant ischemia thought to be a primary contributor to dyspnea
23. Documentation of previous EF < 45%, under stable conditions, within the past 36 months
24. Complex congenital heart disease
25. Uncontrolled hypertension, defined as systolic blood pressure ≥200 mmHg during the screening visit (average value of three blood pressure measurements obtained in supine position)
26. Any other condition that in the judgment of the investigator would jeopardize the patient's participation in the study or that may interfere with the interpretation of study data or if the patient is considered unlikely to comply with study procedures, restrictions and requirements
27. Bariatric surgery within the past 6 months or planned bariatric surgery within the study time course.
28. CardioMems device implantation within previous 4 weeks or planned CardioMems implantation during study period
29. For echo substudy only: patients with ventricular paced rhythm or left bundle branch block on the most recent clinically available 12-lead electrocardiogram.
30. For echo substudy only: permanent atrial fibrillation

Ages: 19 Years to 119 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Kosiborod, MD, Study Chair — Saint Luke's Mid America Heart Institute
Locations (26):
- United States (26):
  - Heart Group of the Eastern Shore, Fairhope, Alabama
  - University of Southern California, Los Angeles, California
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Charlotte Heart Group Research Center, Port Charlotte, Florida
  - Emory University, Atlanta, Georgia
  - NorthShore University HealthSystem Research Insititute, Evanston, Illinois
  - Northwestern University, Evanston, Illinois
  - Chicago Medical Research, Hazel Crest, Illinois
  - OSF HealthCare Cardiovascular Institute, Peoria, Illinois
  - St. Vincent Cardiovascular Research Institute, Indianapolis, Indiana
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Saint Luke's Mid America Heart Institute, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Columbia University, New York, New York
  - St. Francis Hospital, New York, New York
  - Eastern Nephrology Associates, New Bern, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Allegheny Health Network Research Institute, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Scott and White Research Institute, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Eastern Virginia Medical School, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nassif ME, Windsor SL, Borlaug BA, Kitzman DW, Shah SJ, Tang F, Khariton Y, Malik AO, Khumri T, Umpierrez G, Lamba S, Sharma K, Khan SS, Chandra L, Gordon RA, Ryan JJ, Chaudhry SP, Joseph SM, Chow CH, Kanwar MK, Pursley M, Siraj ES, Lewis GD, Clemson BS, Fong M, Kosiborod MN. The SGLT2 inhibitor dapagliflozin in heart failure with preserved ejection fraction: a multicenter randomized trial. Nat Med. 2021 Nov;27(11):1954-1960. doi: 10.1038/s41591-021-01536-x. Epub 2021 Oct 28. PMID 34711976
- [Derived] Selvaraj S, Patel S, Sauer AJ, McGarrah RW, Jones P, Kwee LC, Windsor SL, Ilkayeva O, Muehlbauer MJ, Newgard CB, Borlaug BA, Kitzman DW, Shah SJ, Margulies KB, Husain M, Inzucchi SE, McGuire DK, Lanfear DE, Javaheri A, Umpierrez G, Mentz RJ, Sharma K, Kosiborod MN, Shah SH. Metabolic Effects of the SGLT2 Inhibitor Dapagliflozin in Heart Failure Across the Spectrum of Ejection Fraction. Circ Heart Fail. 2024 Nov;17(11):e011980. doi: 10.1161/CIRCHEARTFAILURE.124.011980. Epub 2024 Oct 18. PMID 39421941
- [Derived] Selvaraj S, Patel S, Sauer AJ, McGarrah RW, Jones P, Kwee LC, Windsor SL, Ilkayeva O, Muehlbauer MJ, Newgard CB, Borlaug BA, Kitzman DW, Shah SJ, Shah SH, Kosiborod MN; PRESERVED-HF Investigators. Targeted Metabolomic Profiling of Dapagliflozin in Heart Failure With Preserved Ejection Fraction: The PRESERVED-HF Trial. JACC Heart Fail. 2024 Jun;12(6):999-1011. doi: 10.1016/j.jchf.2024.02.018. Epub 2024 Apr 17. PMID 38639697
- [Derived] Lewis GD, Gosch K, Cohen LP, Nassif ME, Windsor SL, Borlaug BA, Kitzman DW, Shah SJ, Khumri T, Umpierrez G, Lamba S, Sharma K, Khan SS, Kosiborod MN, Sauer AJ. Effect of Dapagliflozin on 6-Minute Walk Distance in Heart Failure With Preserved Ejection Fraction: PRESERVED-HF. Circ Heart Fail. 2023 Nov;16(11):e010633. doi: 10.1161/CIRCHEARTFAILURE.123.010633. Epub 2023 Oct 23. PMID 37869881
- [Derived] Nassif ME, Windsor SL, Gosch K, Borlaug BA, Husain M, Inzucchi SE, Kitzman DW, McGuire DK, Pitt B, Scirica BM, Shah SJ, Umpierrez G, Austin BA, Lamba S, Khumri T, Sharma K, Kosiborod MN. Dapagliflozin Improves Heart Failure Symptoms and Physical Limitations Across the Full Range of Ejection Fraction: Pooled Patient-Level Analysis From DEFINE-HF and PRESERVED-HF Trials. Circ Heart Fail. 2023 Jul;16(7):e009837. doi: 10.1161/CIRCHEARTFAILURE.122.009837. Epub 2023 May 19. PMID 37203441
- [Derived] Nassif ME, Kosiborod M. Effects of sodium glucose cotransporter type 2 inhibitors on heart failure. Diabetes Obes Metab. 2019 Apr;21 Suppl 2:19-23. doi: 10.1111/dom.13678. PMID 31081589
- See also: Dapagliflozin information — https://druginfo.nlm.nih.gov/drugportal/name/dapagliflozin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dapagliflozin | Placebo
Started | 162 | 162
Completed | 146 | 145
Not Completed | 16 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin | Placebo | Total
Number analyzed (Participants) | 162 | 162 | 324
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69 [64 to 77] | 71 [63 to 78] | 70 [63 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 92 | 184
  Male | 70 | 70 | 140
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 50 | 47 | 97
  White | 108 | 107 | 215
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 162 | 162 | 324
Duration of Heart Failure [Median (Inter-Quartile Range); unit: years] | 3.0 [1.1 to 6.5] | 3.2 [1.0 to 6.6] | 3.0 [1.0 to 6.5]
Previous Hospitalization for Heart Failure [Count of Participants; unit: Participants] | 98 | 83 | 181
Ejection Fraction [Median (Inter-Quartile Range); unit: percent] — Ejection fraction is measured as a percentage of the total amount of blood in the heart that is pumped out with each heartbeat.
  percent | 60 [55 to 65] | 60 [54 to 65] | 60 [55 to 65]
Ischemic Heart Disease [Count of Participants; unit: Participants] | 32 | 31 | 63
Type 2 Diabetes [Count of Participants; unit: Participants] | 90 | 91 | 181
Atrial Fibrillation [Count of Participants; unit: Participants] | 82 | 89 | 171
Internal Cardiac Defibrillator (ICD) [Count of Participants; unit: Participants] | 7 | 9 | 16
Angiotensin converting enzyme inhibitor (ACEI) / Angiotensin II receptor blocker (ARB) [Count of Participants; unit: Participants] | 98 | 98 | 196
Angiotensin receptor-neprilysin inhibitor (ARNI) [Count of Participants; unit: Participants] | 2 | 3 | 5
Beta-blockers [Count of Participants; unit: Participants] | 119 | 116 | 235
Hydralazine [Count of Participants; unit: Participants] | 25 | 18 | 43
Long-Acting Nitrates [Count of Participants; unit: Participants] | 34 | 27 | 61
Mineralocorticoid receptor agonist (MRA) [Count of Participants; unit: Participants] | 50 | 68 | 118
Loop Diuretics [Count of Participants; unit: Participants] | 151 | 135 | 286
Lipid-Lowering Agents [Count of Participants; unit: Participants] | 132 | 127 | 259
Anticoagulant Agents [Count of Participants; unit: Participants] | 71 | 84 | 155
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 35.1 [30.4 to 41.8] | 34.6 [29.7 to 40.4] | 34.7 [30.1 to 41.5]
Heart Rate [Median (Inter-Quartile Range); unit: beats per minute] | 70 [61 to 77] | 68 [62 to 75] | 68 [62 to 76]
Systolic Blood Pressure [Median (Inter-Quartile Range); unit: mm Hg] | 134 [120 to 152] | 132 [118 to 148] | 133 [120 to 149]
N-terminal pro B-type natriuretic peptide (NT-proBNP) - overall [Median (Inter-Quartile Range); unit: pg/mL] | 641 [373 to 1210] | 710 [329 to 1449] | 671 [355 to 1297]
N-terminal pro B-type natriuretic peptide (NT-proBNP) - participants with atrial fibrillation [Median (Inter-Quartile Range); unit: pg/mL] — Population: The number of participants analyzed differs from the overall number of participants analyzed as this analysis has been completed only in participants with a history of atrial fibrillation.
  pg/mL
    number analyzed (Participants) | 82 | 89 | 171
    (all) | 830 [555 to 1711] | 816 [481 to 1687] | 816 [507 to 1693]
N-terminal pro B-type natriuretic peptide (NT-proBNP) - participants with no atrial fibrillation [Median (Inter-Quartile Range); unit: pg/mL] — Population: The number of participants analyzed differs from the overall number of participants analyzed as this analysis has been completed only in participants with no history of atrial fibrillation.
  pg/mL
    number analyzed (Participants) | 80 | 73 | 153
    (all) | 438 [269 to 750] | 485 [263 to 1168] | 459 [266 to 868]
Brain Natriuretic Peptide (BNP) - overall [Median (Inter-Quartile Range); unit: pg/mL] | 137 [81 to 222] | 151 [90 to 254] | 142 [85 to 244]
Brain Natriuretic Peptide (BNP) - participants with atrial fibrillation [Median (Inter-Quartile Range); unit: pg/mL] — Population: The number of participants analyzed differs from the overall number of participants analyzed as this analysis has been completed only in participants with a history of atrial fibrillation.
  pg/mL
    number analyzed (Participants) | 82 | 89 | 171
    (all) | 169 [109 to 255] | 151 [104 to 258] | 154 [107 to 256]
Brain Natriuretic Peptide (BNP) - participants with no atrial fibrillation [Median (Inter-Quartile Range); unit: pg/mL] — Population: The number of participants analyzed differs from the overall number of participants analyzed as this analysis has been completed only in participants with no history of atrial fibrillation.
  pg/mL
    number analyzed (Participants) | 80 | 73 | 153
    (all) | 107 [67 to 179] | 161 [77 to 241] | 128 [71 to 216]
Estimated glomerular filtration rate (eGFR) [Median (Inter-Quartile Range); unit: mL/minute] | 56 [42 to 69] | 54 [41 to 69] | 55 [41 to 69]
Hemoglobin A1c [Median (Inter-Quartile Range); unit: percent of glycosylated hemoglobin] | 6.0 [5.6 to 7.3] | 6.2 [5.6 to 7.1] | 6.1 [5.6 to 7.2]
Hemoglobin [Median (Inter-Quartile Range); unit: g/dL] | 12.7 [11.5 to 13.9] | 12.6 [11.6 to 13.8] | 12.6 [11.5 to 13.9]
New York Heart Association (NYHA) Class II [Count of Participants; unit: Participants] — NYHA Functional Classification places patients in one of four categories based on how much they are limited during physical activity. A higher class means a worse functional condition. NYHA Class II indicates the patient has been classified as having slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  Participants | 96 | 90 | 186
New York Heart Association (NYHA) Class III/IV [Count of Participants; unit: Participants] — NYHA Functional Classification places patients in one of four categories based on how much they are limited during physical activity A higher class means a worse functional condition. NYHA Class III indicates the patient has been classified as having marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea. NYHA Class IV indicates the patient has been classified Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
  Participants | 65 | 72 | 137
Kansas City Cardiomyopathy Questionnaire - Overall Summary Score (KCCQ-OS) [Mean (Standard Deviation); unit: units on a scale] — The KCCQ is a disease-specific health status instrument composed of 23 items that quantifies the domains of physical limitations, symptoms, self-efficacy, social limitation and quality of life from heart failure. Scores range from 0-100, in which higher scores reflect better health status.
  units on a scale | 63.2 (20.4) | 62.3 (20.6) | 62.7 (20.4)
Kansas City Cardiomyopathy Questionnaire - Clinical Summary Score (KCCQ-CS) [Mean (Standard Deviation); unit: units on a scale] — The KCCQ is a disease-specific health status instrument composed of 23 items that quantifies the domains of physical limitations, symptoms, self-efficacy, social limitation and quality of life from heart failure. Scores range from 0-100, in which higher scores reflect better health status.
  units on a scale | 63.4 (19.7) | 61.8 (20.3) | 62.6 (20.0)
6 minute walk test [Median (Inter-Quartile Range); unit: meters] | 244 [165 to 329] | 244 [154 to 317] | 244 [162 to 326]

OUTCOME MEASURES:

1. Primary Outcome: Effect of Dapagliflozin, as Compared With Placebo, on Heart Failure Related Health Status Using the Kansas City Cardiomyopathy Questionnaire Clinical Summary Summary Score (KCCQ-CS)
Description: Kansas City Cardiomyopathy Questionnaire clinical summary score (KCCQ-CS) at Week 12.
  The KCCQ is a disease-specific health status instrument composed of 23 items that quantifies the domains of physical limitations, symptoms, self-efficacy, social limitation and quality of life from heart failure. Scores range from 0-100, in which higher scores reflect better health status. For the KCCQ-CS, a small but clinically meaningful change is considered to be ≥ 5 points.
  Values have been adjusted for the corresponding baseline value, history of type 2 diabetes, sex, atrial fibrillation, baseline estimated glomerular filtration rate and left ventricular ejection fraction.
Time Frame: Baseline to Week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 162 | 162
score on a scale | 68.6 [66.2 to 71.0] | 62.8 [60.4 to 65.3]

2. Secondary Outcome: Effect of Dapagliflozin, as Compared With Placebo, on Heart Failure Related Health Status Using the Kansas City Cardiomyopathy Questionnaire Overall Summary Score (KCCQ-OS)
Description: Kansas City Cardiomyopathy Questionnaire overall summary score (KCCQ-OS) at Week 12.
  The KCCQ is a disease-specific health status instrument composed of 23 items that quantifies the domains of physical limitations, symptoms, self-efficacy, social limitation and quality of life from heart failure. Scores range from 0-100, in which higher scores reflect better health status. For the KCCQ-OS, a small but clinically meaningful change is considered to be ≥ 5 points.
  Values have been adjusted for the corresponding baseline value, history of type 2 diabetes, sex, atrial fibrillation, baseline estimated glomerular filtration rate and left ventricular ejection fraction.
Time Frame: Baseline to Week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 162 | 162
score on a scale | 68.9 [66.5 to 71.3] | 64.5 [62.1 to 66.8]

3. Secondary Outcome: Effect of Dapagliflozin, as Compared With Placebo, on N-terminal Pro B-type Natriuretic Peptide (NTproBNP)
Description: NTproBNP at Week 12. Values have been adjusted for the corresponding baseline value, history of type 2 diabetes, sex, atrial fibrillation, baseline estimated glomerular filtration rate and left ventricular ejection fraction.
Time Frame: Baseline to Week 12
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 162 | 162
pg/mL | 733 [673 to 799] | 739 [678 to 805]

4. Secondary Outcome: Effect of Dapagliflozin, as Compared With Placebo, on Brain Natriuretic Peptide (BNP)
Description: BNP at Week 12. Values have been adjusted for the corresponding baseline value, history of type 2 diabetes, sex, atrial fibrillation, baseline estimated glomerular filtration rate and left ventricular ejection fraction.
Time Frame: Baseline to Week 12
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 162 | 162
pg/mL | 147 [136 to 160] | 147 [136 to 160]

5. Secondary Outcome: Effect of Dapagliflozin, as Compared With Placebo, on 6 Minute Walk Test Distance
Description: 6 minute walk test distance at 12 weeks. Values have been adjusted for the corresponding baseline value, history of type 2 diabetes, sex, atrial fibrillation, baseline estimated glomerular filtration rate and left ventricular ejection fraction.
Time Frame: Baseline to Week 12
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 162 | 162
meters | 262 [252 to 272] | 242 [232 to 252]

6. Secondary Outcome: Effect of Dapagliflozin, as Compared With Placebo, on Hemoglobin A1c
Description: Hemoglobin A1c at Week 12. Values have been adjusted for the corresponding baseline value, history of type 2 diabetes, sex, atrial fibrillation, baseline estimated glomerular filtration rate and left ventricular ejection fraction.
Time Frame: Baseline to Week 12
Measure: Mean (95% Confidence Interval); unit: Percent
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 162 | 162
Percent | 6.5 [6.4 to 6.6] | 6.6 [6.5 to 6.7]

7. Secondary Outcome: Effect of Dapagliflozin, as Compared With Placebo, on the Proportion of Patients With a ≥ 5 Point Increase in KCCQ Clinical Summary Score (KCCQ-CS) and KCCQ Overall Summary Score (KCCQ-OS)
Description: Proportion of patients with a ≥ 5 point increase in KCCQ-CS and KCCQ-OS at Week 12.
  The KCCQ is a disease-specific health status instrument composed of 23 items that quantifies the domains of physical limitations, symptoms, self-efficacy, social limitation and quality of life from heart failure. Scores range from 0-100, in which higher scores reflect better health status. For KCCQ-CS and KCCQ-OS, a small but clinically meaningful change is considered to be ≥ 5 points.
  Values have been adjusted for the corresponding baseline value, history of type 2 diabetes, sex, atrial fibrillation, baseline estimated glomerular filtration rate and left ventricular ejection fraction.
Time Frame: Baseline to Week 12
Population: The number of participants analyzed may differ from the overall number of participants analyzed due to missing data at certain timepoints for some participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 152 | 152
Participants
  KCCQ-CS increase ≥ 5 points | 69 | 53
  KCCQ-OS increase ≥ 5 points | 75 | 58

8. Secondary Outcome: Effect of Dapagliflozin, as Compared With Placebo, on the Proportion of Patients With a ≥ 20% Decrease in N-terminal Pro B-type Natriuretic Peptide (NTproBNP)
Description: Proportion of patients with a ≥ 20% decrease in NTproBNP at Week 12. Values have been adjusted for the corresponding baseline value, history of type 2 diabetes, sex, atrial fibrillation, baseline estimated glomerular filtration rate and left ventricular ejection fraction.
Time Frame: Baseline to Week 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 150 | 150
Participants | 48 | 44

9. Secondary Outcome: Effect of Dapagliflozin, as Compared With Placebo, on Proportion of Patients With ≥ 5 Point Increase in Kansas City Cardiomyopathy Questionnaire Clinical Summary Score (KCCQ-CS) and ≥ 20% Decrease in N-terminal Pro B-type Natriuretic Peptide(NTproBNP)
Description: Proportion of patients with a ≥ 5 point increase in KCCQ-CS and a ≥ 20% decrease in NTproBNP at Week 12. Values have been adjusted for the corresponding baseline value, history of type 2 diabetes, sex, atrial fibrillation, baseline estimated glomerular filtration rate and left ventricular ejection fraction.
Time Frame: Baseline to Week 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 148 | 150
Participants | 23 | 15

10. Secondary Outcome: Effect of Dapagliflozin, as Compared With Placebo, on Weight
Description: Weight at Week 12. Values have been adjusted for the corresponding baseline value, history of type 2 diabetes, sex, atrial fibrillation, baseline estimated glomerular filtration rate and left ventricular ejection fraction.
Time Frame: Baseline to Week 12
Measure: Mean (95% Confidence Interval); unit: kilograms
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 162 | 162
kilograms | 101.3 [100.9 to 101.8] | 102.1 [101.6 to 102.6]

11. Secondary Outcome: Effect of Dapagliflozin, as Compared With Placebo, on Systolic Blood Pressure
Description: Systolic blood pressure at Week 12. Values have been adjusted for the corresponding baseline value, history of type 2 diabetes, sex, atrial fibrillation, baseline estimated glomerular filtration rate and left ventricular ejection fraction.
Time Frame: Baseline to Week 12
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 162 | 162
mm Hg | 133 [130 to 135] | 133 [131 to 136]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for up to 15 weeks. The adverse event collection period started at the time the patient signed consent at their Screening Visit, continued through a 12-week double-blind treatment period after randomization, and ended after completion of a 1-week follow-up period after completion of the double-blind treatment period.
Description: Serious Adverse Events, Drug Adverse Events, Adverse Events of Special Interest and Urgent Outpatient Heart Failure Visits were collected. A Drug Adverse Event is an adverse event which leads to premature and permanent discontinuation of study medication. Adverse Events of Special Interest include diabetic ketoacidosis, volume depletion (defined as hypotension, syncope, orthostatic hypotension or dehydration), severe hypoglycemic events and lower limb amputations.
Arm/Group | Dapagliflozin | Placebo
All-Cause Mortality (participants affected / at risk) | 1/162 | 2/162
Serious Adverse Events (participants affected / at risk) | 31/162 | 22/162
Other Adverse Events (participants affected / at risk) | 13/162 | 16/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin (N=162) | Placebo (N=162)
Abdominal Wall Hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acute Kidney Injury (General disorders) | 8 (8) | 4 (4)
Acute Renal Failure (General disorders) | 1 (1) | 0 (0)
Acute Respiratory Distress (General disorders) | 1 (1) | 0 (0)
Acute Right Cerebellar Infarct (General disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ascites of the Abdomen (Hepatobiliary disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 3 (3) | 0 (0)
Atrial Flutter (Cardiac disorders) | 1 (1) | 1 (1)
Benign Paroxysmal Positional Vertigo (General disorders) | 1 (1) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 3 (3)
Chest Pain (General disorders) | 0 (0) | 2 (2)
Clostridium Difficile (Infections and infestations) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 2 (2)
Critical Limb Ischemia (General disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Elective Watchman Device Implantation (Cardiac disorders) | 0 (0) | 1 (1)
Elevated Troponin in the setting of Covid-19 (General disorders) | 1 (1) | 0 (0)
Exacerbation of Chronic Obstructive Pulmonary Disease (General disorders) | 0 (0) | 1 (1)
Exacerbation of Heart Failure (Cardiac disorders) | 14 (17) | 6 (7)
Gastroenteritis (Eye disorders) | 1 (1) | 0 (0)
Gastrointestinal bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hematuria (General disorders) | 0 (0) | 1 (1)
Hemochromatosis (General disorders) | 1 (1) | 0 (0)
Hemoptysis (General disorders) | 1 (1) | 0 (0)
Hypercapnic and hypoxic respiratory failure requiring intubation (General disorders) | 1 (1) | 0 (0)
Hyperglycemia (General disorders) | 1 (1) | 1 (1)
Hypotension (General disorders) | 1 (1) | 0 (0)
Infected right great toe (Infections and infestations) | 0 (0) | 1 (1)
Influenza A (Infections and infestations) | 0 (0) | 1 (1)
Iron Overload cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Left hilar mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Left hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Liver failure/Cirrhosis leading to Hepatic/Metabolic Encephalopathy (Hepatobiliary disorders) | 0 (0) | 1 (1)
Melena and hematochezia (General disorders) | 1 (1) | 0 (0)
Multiple Abscesses (Infections and infestations) | 0 (0) | 1 (1)
Non cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Osteoarthritis (Right Hip) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteomyelitis (left foot) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Parainfluenza (Infections and infestations) | 1 (1) | 0 (0)
Aortic Ulcer (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal failure leading to endstage renal disease requiring dialysis (General disorders) | 0 (0) | 1 (1)
Right leg pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Right Shoulder - Infected Arthroplasty (Infections and infestations) | 1 (1) | 0 (0)
Salmonella enteritis/diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Schwannoma of spinal cord at L1-L2 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Septic Arthritis of the Right Knee (Infections and infestations) | 0 (0) | 1 (1)
Septicemia (Infections and infestations) | 1 (1) | 0 (0)
Endstage chronic obstructive pulmonary disease with hypoxic and hypercapnic respiratory failure (General disorders) | 0 (0) | 1 (1)
Suicidal Ideation (General disorders) | 2 (2) | 0 (0)
Syncope (General disorders) | 1 (1) | 0 (0)
Type II NSTEMI (Cardiac disorders) | 1 (1) | 0 (0)
Uncontrolled Hypertension (General disorders) | 1 (1) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Volume Depletion (General disorders) | 2 (2) | 1 (2)
Hypertensive Crisis (General disorders) | 1 (1) | 0 (0)
Worsening Osteoarthritis - Left Knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin (N=162) | Placebo (N=162)
Volume Depletion (General disorders) | 10 (11) | 7 (7)
Urgent Heart Failure Visit (Cardiac disorders) | 8 (8) | 8 (13)
Nausea (General disorders) | 1 (1) | 0 (0)
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal intolerance (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary frequency (General disorders) | 1 (1) | 0 (0)
Rash (General disorders) | 0 (0) | 1 (1)
Blurry vision (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Shortness of Breath (General disorders) | 0 (0) | 1 (1)
Foul smelling urine (General disorders) | 1 (1) | 0 (0)
Sense of hopelessness (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor will have 18 months after the study closure to arrange for the submission of multicenter publications. If multicenter publications are not submitted within 24 months after conclusion of the study, PI may publish the results from their site's data, pursuant to approval by the Sponsor and Executive Committee at least 60 days prior to submission. The Sponsor cannot require changes to the communication with the exception of requiring the removal of confidential information.

DOCUMENTS (2):
  • Study Protocol (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT03030235/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/35/NCT03030235/SAP_001.pdf